CLINICAL TRIAL: NCT05161169
Title: Implementation of Whole Genome Sequencing as Screening in a Diverse Cohort of Healthy Infants (1U01TR003201-01A1)
Brief Title: Implementation of Whole Genome Sequencing as Screening in a Diverse Cohort of Healthy Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Baylor College of Medicine (Other); Boston Children's Hospital (Other); Broad Institute of MIT and Harvard (Other); Dartmouth-Hitchcock Medical Center (Other); Harvard Pilgrim Health Care (Other); Howard University (Other); HudsonAlpha Institute for Biotechnology (Other); Massachusetts General Hospital (Other); Icahn School of Medicine at Mount Sinai (Other); University of Alabama at Birmingham (Other); National Center for Advancing Translational Sciences (NCATS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Robert C. Green, MD, MPH, Professor of Medicine (Genetics), Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: The BabySeq2 Project
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Genetic Predisposition to Disease; Hereditary Diseases
Keywords: genome sequencing; newborn screening; preventive medicine
MeSH Terms: conditions — Genetic Predisposition to Disease; Genetic Diseases, Inborn

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (control group vs. genome sequencing intervention)
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequencing cohort (Experimental): Infants receive genome sequencing with analysis of approximately 1000 genes associated with childhood-onset and highly actionable adult-onset disease risks. Pathogenic and likely pathogenic variants are reported to the child's parents and pediatrician. Participants also receive a detailed family history report and standard well-child care.
  Interventions: Genetic: Genome Sequencing
- Control cohort (No Intervention): Infants receive a detailed family history report plus standard well-child care.

INTERVENTIONS:
Genetic: Genome Sequencing — 20 times read depth (20x) next-generation whole genome sequencing with comprehensive analysis.
  Arms: Sequencing cohort

SUMMARY:
This research study is exploring the use of genomic sequencing in the newborn period to screen healthy babies for current and future health risks. The study will enroll a diverse cohort of 500 healthy infants and their parents from Boston, MA; New York City, NY; and Birmingham, AL. A small blood sample will be collected from each infant, and whole genome sequencing will be performed in 1/2 of the cohort following a randomized controlled trial design. 3 months later, the randomization status and sequencing results will be shared with parents and pediatricians. Investigators will study the medical, behavioral, and economic outcomes of genomic sequencing to better understand how this technology can be implemented in outpatient primary care settings.

DETAILED DESCRIPTION:
The objective of this research protocol is to assess the impacts of genomic sequencing in healthy infants from ethnically and racially diverse communities as part of routine pediatric care.

Investigators will enroll a cohort of 500 healthy, ethnically and racially diverse infants from Boston, Massachusetts; New York City, New York; and Birmingham, Alabama, with planned expansion to other U.S. cities and recruitment sites. As part of this study, a stakeholder board comprised of diverse community members will provide early and regular feedback throughout the study on anticipated and ongoing community reaction to the work with sensitivity to historical injustices and cultural diversity

Primary care pediatricians from each recruitment site will be enrolled for a brief genomics education curriculum. Only infants whose healthcare providers have joined the study will be enrolled.

A small blood sample will be obtained from each enrolled infant. Participants will randomized (1:1) to receive either a family history report or a family history report plus whole genome sequencing.

Genome sequencing data will be analyzed for pathogenic and likely pathogenic variants in genes associated with childhood-onset disease risks, as well as highly actionable adult-onset disease risks. If infants have a dominant risk identified, parents may choose to be screened as part of the study.

The study team will disclose the infant's randomization status and study results during a consultation with each family, and results will be sent to the infant's pediatrician.

Parents will be surveyed at three time points over the 12 months after enrollment: baseline, immediately post-disclosure (approximately 3 months after enrollment), and 6 months post-disclosure. Surveys will assess psychosocial impacts of newborn sequencing.

Chart reviews will be performed to assess the medical outcomes and healthcare utilization costs of newborn genome sequencing.

ELIGIBILITY:
Inclusion Criteria:

Infant participants

* Has not previously had exome or genome sequencing
* Age 0-12 months
* Seen for well-baby pediatric care at a recruiting site
* Primary healthcare provider completed the genomics education program
* At least one parent or guardian able to participate in the study

Parent participants

* Biological parent or legal guardian of an infant participating in the study
* 18 years of age or older
* Unimpaired decision-making capacity
* English or Spanish speaking
* Available to have genetic counseling and provide consent for testing the infant

Exclusion Criteria:

* Parents are unwilling to have genomic reports placed in the medical record or sent to their primary care pediatrician
* Any infant in which clinical considerations preclude collecting blood via heel stick

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Monogenic disease risks (MDRs) | 3 months after enrollment
  Pathogenic (P) and likely pathogenic (LP) variants identified relevant to infant's health (dominant or biallelic recessive disease risks)
Carrier status variants | 3 months after enrollment
  P and LP variants identified as recessive carrier status in infant
MDR-associated phenotype | 3 months after enrollment and 1-year post-disclosure (15 months after enrollment)
  Signs or symptoms of monogenic disease risk identified by genome sequencing
Parenting stress, relationship dysfunction | Baseline, post-disclosure (3 months after enrollment), 6 months post-disclosure (9 months after enrollment)
  Parenting Stress Index, 4th Edition Short Form (scored as a percentile 0 - 100%, higher scores indicate increased stress)
Relationship satisfaction | Baseline, post-disclosure (3 months after enrollment), 6 months post-disclosure (9 months after enrollment)
  Kansas Marital Satisfaction Scale (Scored 3 to 21, higher scores indicate better marital quality)
General anxiety | Baseline, post-disclosure (3 months after enrollment), 6 months post-disclosure (9 months after enrollment)
  General Anxiety Disorder-7

SECONDARY OUTCOMES:
MDR-associated family history | 3 months after enrollment and 1-year post-disclosure (15 months after enrollment)
  Signs or symptoms of monogenic disease risk or recessive condition present in infant's biological family
Intervention prompted by genetic or family history report | 6 months post-disclosure (9 months after enrollment)
  Healthcare intervention prompted by MDR or recessive carrier variant
Suspected genetic condition | 6 months post-disclosure (9 months after enrollment)
  Any phenotype that develops in an infant or a family history suspected to have a genetic cause
Child vulnerability | Baseline, post-disclosure (3 months after enrollment), 6 months post-disclosure (9 months after enrollment)
  Vulnerable Baby Scale (scored 0-50, higher scores indicate increased perceptions of child vulnerability)
Feelings about genomic testing | Baseline, post-disclosure (3 months after enrollment), 6 months post-disclosure (9 months after enrollment)
  Feelings About genomiC Testing Results (FACToR) Questionnaire
Partner blame | Baseline, post-disclosure (3 months after enrollment), 6 months post-disclosure (9 months after enrollment)
  Novel item (higher scores indicate increased blame)
General depression | Baseline, post-disclosure (3 months after enrollment), 6 months post-disclosure (9 months after enrollment)
  Patient Health Questionnaire (PHQ)-8
Self blame | Baseline, post-disclosure (3 months after enrollment), 6 months post-disclosure (9 months after enrollment)
  Novel item (higher scores indicate increased blame)

OTHER OUTCOMES:
Cost of attributable services | 6 months post-disclosure (9 months after enrollment)
  Cost of health care services associated with surveillance and diagnosis of GS and family history risks
Cost of genomic services | 6 months post-disclosure (9 months after enrollment)
  Cost of genetic services infants and parents received after study disclosure session
All healthcare costs | 6 months post-disclosure (9 months after enrollment)
  All health sector costs observed in medical records and survey questions regarding family out-of-pocket expenses

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Green, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Ingrid A. Holm, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Boston Children's Hospital, Boston, Massachusetts
  - Beaumont - Corewell Health East, Royal Oak, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and statistical analysis plan will be shared on clinical trials.gov
Supporting Information: Study Protocol, SAP
Time Frame: Supporting information will be shared 6 months after study completion.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT05161169/Prot_SAP_000.pdf